CLINICAL TRIAL: NCT05544682
Title: Cefiderocol in the Treatment of Multidrug-resistant Gram-negative Bacilli Infections, a Retrospective Study
Acronym: CefiNoFer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8701
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Multidrug Resistant Bacterial Infection
Keywords: Multidrug Resistant Bacterial Infections; Gram-negative bacilli infections; Cefiderocol; Antibiotics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cefiderocol is a new antibiotic from the siderophore cephalosporin family for which there are few real-life data on its use in the treatment of infections with multidrug-resistant Gram-negative bacilli.

The circulation of bacterial strains multi-resistant to antibiotics is important at the Strasbourg University Hospital, so the investigators wish to report their local experience of the 1st uses of Cefiderocol in the treatment of infections with multi-resistant Gram-negative bacilli to antibiotics in order to better clarify the use of this antibiotic (therapeutic indication, method of administration)

ELIGIBILITY:
Inclusion criteria:

* Adult patient (≥18 years old)
* taken care of in the HUS and treated as part of routine care with Cefiderocol between 04/01/2020 and 08/31/2022.
* Subjects who have not expressed their opposition to the reuse of their data for scientific research purposes.

Exclusion criteria:

- Patient who has expressed his opposition to the retrospective reuse of his data for scientific research purposes.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient (≥18 years old) taken care of in the HUS and treated as part of routine care with Cefiderocol between 04/01/2020 and 08/31/2022.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Retrospective evaluation of the therapeutic management of patients treated as part of routine care with Cefiderocol | 30 days post treatment with Céfiderocol
  Survival, significant clinical improvement, absence of microbiological failure or infectious recurrence on day 30 after treatment with Céfiderocol

CONTACTS AND LOCATIONS:
Locations (1):
- Service des maladies infectieuses et tropicales - CHU de Strasbourg - France, Strasbourg, France